CLINICAL TRIAL: NCT01597856
Title: Evaluation and Treatment of Substance Use in Veterans With PTSD Disability Claims
Brief Title: Evaluation and Treatment of Substance Abuse in Veterans With PTSD Disability Claims
Acronym: SBIRT-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 11-091
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Attendance at Treatment; PTSD, Substance Use, and Attendance at Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBIRT (Experimental): The SBIRT-VA manual codifies basic substance abuse screening, treatment, Motivational Interviewing and referral procedures. It is designed for providers with minimal substance abuse expertise and is easy for experienced substance abuse providers to deliver.
  Study sessions include identifying the Veterans' values through a card sort, the change ruler, on which the Veteran rates his/her willingness to change current behavior, listing the pros and cons of changing.
  Interventions: Behavioral: SBIRT
- No additional treatment (No Intervention): Veterans assigned to the control condition will not receive any study-related therapy. A Veteran who completes a Compensation examination ordinarily has no further treatment, referral, or debriefing as part of the Compensation examination.

INTERVENTIONS:
Behavioral: SBIRT — SBIRT Therapy overview-
  1. Therapist explains purpose of the therapy.
  2. Inquiry about Compensation examination-ask if Veteran has questions about determination process and address concerns.
  3. Discuss relationship between PTSD and substance use- long-term substance use is a form of avoidance and barrier to recovery.
  4. Discuss treatment needs, administer screening, provide feedback.
  Arms: SBIRT

SUMMARY:
Veterans can apply for compensation and pension (C & P) benefits for a disability related to military service. The application exam for these benefits provides an opportunity for Veterans returning from service to access VA care. The investigators will recruit Veterans applying for C & P to participate in this study. All enrolled participants will complete questionnaires around the time of their C & P exam related to substance abuse, PTSD, service use, and attitudes. The investigators will monitor enrolled Veterans' attendance at treatment over time, and examine whether C & P award, substance use, and beliefs about benefits are related to treatment attendance. Some enrolled participants will be assigned to one of two study groups: a treatment group and a no-additional-treatment group. People assigned to these groups will complete the same substance abuse, PTSD, service use, and attitudes questionnaires two additional times during the study. Participants assigned to the treatment group will receive information about the relationship between substance use and PTSD and will be referred to relevant treatment. The investigators will test whether Veterans who receive no-additional-treatment have different symptoms over time and attend less treatment sessions (mental health or substance abuse) than people assigned to treatment.

DETAILED DESCRIPTION:
The Compensation examination that determines if a Veteran is entitled to any disability payments related to military service is a crucial gateway to accessing VA care for returning OEF/OIF Veterans. However, researchers and oversight agencies have noted that examiners typically do not have guidelines for evaluating comorbid conditions like substance abuse and for referring patients to treatment.

In the Evaluative Component of this study, OEF/OIF Veterans presenting for Compensation evaluations for PTSD will be approached to undergo a paid battery of confidential substance use, PTSD, service use and attitude assessments prior to their scheduled Compensation examinations. The batteries will be collected again twice, four and twelve weeks after the Compensation examinations. Long-term follow-up data will be extracted from VA databases including diagnoses, the results of the Veterans' Compensation evaluations, award determination, use of VA services and attendance at mental health and/or substance abuse treatment.

In the Clinical Trial Component of this study, one hundred sixty Veterans identified during the baseline evaluation as having a substance use disorder will be randomly assigned to a session of Screening, Brief Intervention and Referral to Treatment (SBIRT) or to No-Additional-Treatment. SBIRT is an approach to identifying and treating patients with substance abuse issues who are presenting for purposes other than substance abuse treatment. It involves Motivational Interviewing, which has been a consistently effective approach to facilitating engagement in substance abuse treatment in Veterans (Davis, Baer et al. 2003) and other populations. The study will examine factors associated with attendance at treatment including substance use, Veterans' beliefs about benefits, and compensation award. Group comparisons will be conducted on rates of treatment attendance, alcohol use, and PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of OEF or OIF,
* Not currently receiving VBA Compensation for PTSD,
* Able to participate psychologically and physically, able to give informed consent and complete, assessments, and participate in study procedures
* Between the ages of 18-65 years old.

Exclusion Criteria:

* Will not be able to attend the week 4 or 12 appointment because of anticipated incarceration or move

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jankowski RL, Black AC, Lazar CM, Brummett BR, Rosen MI. Consideration of substance use in compensation and pension examinations of veterans filing PTSD claims. PLoS One. 2019 Feb 6;14(2):e0210938. doi: 10.1371/journal.pone.0210938. eCollection 2019. PMID 30726261
- [Result] Black AC, Meshberg-Cohen S, Perez-Ortiz AC, Thornhill TA, Rosen MI. Veterans' compensation claims beliefs predict timing of PTSD treatment use relative to compensation and pension exam. PLoS One. 2018 Dec 27;13(12):e0209488. doi: 10.1371/journal.pone.0209488. eCollection 2018. PMID 30589882
- [Result] Meshberg-Cohen S, Kachadourian L, Black AC, Rosen MI. Relationship between substance use and attitudes towards seeking professional psychological help among veterans filing PTSD claims. Addict Behav. 2017 Nov;74:9-12. doi: 10.1016/j.addbeh.2017.05.024. Epub 2017 May 23. PMID 28558337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post 9-11 era Veterans with an initial PTSD Compensation & Pension Application scheduled were recruited from VA Connecticut Healthcare System and TN Valley Healthcare system between April 2013 and July 2016.
Pre-assignment Details: All enrolled Veterans completed study assessments at baseline, week 4 and week 12. Only Veterans with self-reported risky alcohol use or use of an illicit drug within the last 28 days were randomized to receive SBIRT counseling or No additional counseling conditions.
Groups:
- SBIRT: The SBIRT-VA manual codifies basic substance abuse screening, treatment, Motivational Interviewing and referral procedures. It is designed for providers with minimal substance abuse expertise and is easy for experienced substance abuse providers to deliver.
  Study sessions include identifying the Veterans' values through a card sort, the change ruler, on which the Veteran rates his/her willingness to change current behavior, listing the pros and cons of changing.
  SBIRT: SBIRT Therapy overview-
  1. Therapist explains purpose of the therapy.
  2. Inquiry about Compensation examination-ask if Veteran has questions about determination process and address concerns.
  3. Discuss relationship between PTSD and substance use- long-term substance use is a form of avoidance and barrier to recovery.
  4. Discuss treatment needs, administer screening, provide feedback.
- Not Randomized: Enrolled Veterans with no risky substance use.
Period: Overall Study
Arm/Group | SBIRT | No Additional Treatment | Not Randomized
Started | 85 | 87 | 174
Week 4 Follow-up | 62 | 67 | 129
Completed | 63 | 61 | 120
Not Completed | 22 | 26 | 54

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Veterans enrolled who did not report risky substance use at baseline.
- Total: Total of all reporting groups
Arm/Group | SBIRT | No Additional Treatment | Not Randomized | Total
Number analyzed (Participants) | 85 | 87 | 174 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (7.8) | 32.4 (7.6) | 36.6 (9.6) | 34.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 24 | 46
  Male | 70 | 80 | 150 | 300
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 3 | 6
  Black (not Hispanic) | 15 | 14 | 32 | 61
  White (not Hispanic) | 55 | 60 | 112 | 227
  Hispanic | 10 | 8 | 24 | 42
  Other | 3 | 4 | 3 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 87 | 174 | 346

OUTCOME MEASURES:

1. Primary Outcome: Treatment Attendance by Treatment Group Over Time
Description: Mean number of weeks of substance abuse and/or mental health treatment attended (as measured by the Electronic Medical Record) by treatment group over time
Time Frame: 4 weeks pre-baseline through week 12 post baseline, total of 16 Weeks
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- SBIRT: Intervention Group
- No Additional Treatment: Control Group (Randomized, no intervention)
- Not Randomized: Comparison Group (no risky substance use at baseline)
Arm/Group | SBIRT | No Additional Treatment | Not Randomized
Number analyzed (Participants) | 85 | 87 | 174
weeks
  4 weeks Pre-Baseline | 0.75 (1.18) | 0.53 (0.92) | 0.83 (1.20)
  Baseline to week 4 | 0.89 (1.22) | 0.55 (0.81) | 0.94 (1.16)
  Week 4 to week 12 | 1.98 (2.19) | 0.98 (1.50) | 1.71 (2.30)

2. Secondary Outcome: Substance Use by Treatment Group Over Time
Description: Mean days self-reported risky drug or alcohol use
Time Frame: 4 weeks pre-baseline through week 12 post baseline, total of 16 Weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SBIRT | No Additional Treatment | Not Randomized
Number analyzed (Participants) | 85 | 87 | 174
days
  4 weeks Pre-Baseline | 2.12 (1.67) | 2.39 (1.66) | 0.98 (1.53)
  Baseline to Week 4 | 1.73 (1.83) | 1.63 (1.80) | 0.98 (1.50)
  Week 4 to Week 12 | 2.60 (3.24) | 2.77 (3.18) | 1.80 (2.80)

3. Secondary Outcome: Mean PTSD Severity Score
Description: Measure on Clinical Assessment of PTSD Severity (CAPS IV) rating scale (range 0-136, higher is more severe symptoms).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBIRT | No Additional Treatment | Not Randomized
Number analyzed (Participants) | 85 | 87 | 174
score on a scale
  Baseline | 63.13 (20.74) | 59.63 (22.42) | 59.98 (21.95)
  Week 4 | 58.54 (20.68) | 49.69 (22.23) | 54.34 (24.13)
  Week 12 | 55.24 (23.88) | 48.96 (23.34) | 52.17 (22.42)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Not Randomized: Veterans reporting no risky substance use at baseline.
Arm/Group | SBIRT | No Additional Treatment | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/87 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/87 | 0/174
Other Adverse Events (participants affected / at risk) | 0/85 | 0/87 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT01597856/Prot_SAP_000.pdf